CLINICAL TRIAL: NCT06913192
Title: A Single-Center, Open-Label, Single-Arm Clinical Study of Sequential Anti-BCMA CAR-T Cell Therapy Following Autologous Hematopoietic Stem Cell Transplantation in Transplant-Eligible Newly Diagnosed Multiple Myeloma
Brief Title: Efficacy of Sequential BCMA CAR-T Cell Therapy Following Autologous Hematopoietic Stem Cell Transplantation in Transplant-eligible Newly Diagnosed Multiple Myeloma
Acronym: AUTO-CAR-T
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Pro., Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2025-KL063-01; XYFY2025-KL063-01 (Other: The Affiliated Hospital oh Xuzhou Medical University)
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T following ASCT (Experimental): All enrolled patients will receive three cycles of induction therapy using either the DVRd regimen (Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone) or the DKRd regimen (Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone). Following induction, patients will undergo high-dose melphalan conditioning followed by autologous hematopoietic stem cell transplantation. On Day 5 after stem cell reinfusion, patients will receive anti-BCMA CAR-T cell infusion. After CAR-T therapy, patients will enter the maintenance phase with lenalidomide monotherapy or lenalidomide in combination with bortezomib until disease progression or intolerable toxicity occurs.
  Interventions: Biological: CAR-T

INTERVENTIONS:
Biological: CAR-T — All enrolled patients will receive three cycles of induction therapy using either the DVRd regimen (Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone) or the DKRd regimen (Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone). Following induction, patients will undergo high-dose melphalan conditioning followed by autologous hematopoietic stem cell transplantation. On Day 5 after stem cell reinfusion, patients will receive anti-BCMA CAR-T cell infusion. After CAR-T therapy, patients will enter the maintenance phase with lenalidomide monotherapy or lenalidomide in combination with bortezomib until disease progression or intolerable toxicity occurs.

SUMMARY:
1. Study Title A Single-Center, Open-Label, Single-Arm Clinical Study of Sequential Anti-BCMA CAR-T Cell Therapy Following Autologous Hematopoietic Stem Cell Transplantation in Transplant-Eligible Newly Diagnosed Multiple Myeloma
2. Study Objective This study aims to evaluate the safety and efficacy of sequential anti-BCMA CAR-T cell therapy following autologous hematopoietic stem cell transplantation (ASCT) in transplant-eligible patients with newly diagnosed multiple myeloma (NDMM), in order to provide evidence for optimizing treatment strategies in this population.
3. Study Design This is a single-center, open-label, single-arm clinical study. A total of 50 patients with newly diagnosed multiple myeloma who meet the inclusion criteria will be enrolled. All participants will receive a standardized treatment regimen and undergo regular follow-up for efficacy and safety assessments.
4. Study Population and Eligibility Criteria (1) Inclusion Criteria Age between 18 and 70 years;

Estimated life expectancy > 12 weeks;

Diagnosis of multiple myeloma confirmed by physical examination, histopathology, laboratory tests, and imaging;

Liver function: ALT and AST < 3 times the upper limit of normal;

Karnofsky Performance Status (KPS) score > 50%;

No severe dysfunction of major organs such as the liver or heart;

Willingness to undergo ASCT and CAR-T cell therapy for multiple myeloma;

Ability to provide peripheral venous blood and no contraindications to leukapheresis;

Ability to understand the study and sign a written informed consent voluntarily.

(2) Exclusion Criteria Pregnant or lactating women, or those planning pregnancy within six months;

Patients with infectious diseases, including HIV infection or active tuberculosis;

Patients with active hepatitis B or C virus infection;

Pre-screening indicates peripheral blood T cell transduction efficiency <10% or expansion fold <5× under CD3/CD28 co-stimulation;

Patients with abnormal vital signs or unable to cooperate with the procedures;

Patients with psychiatric or psychological disorders that impair compliance or assessment;

Patients with a history of severe allergies or hypersensitivity, particularly to interleukin-2 (IL-2);

Patients with systemic or severe local infections requiring anti-infective therapy;

Patients with significant dysfunction of vital organs such as the heart, lungs, or brain;

Any other condition deemed unsuitable for participation by the investigator.

5. Treatment Protocol All enrolled patients will receive three cycles of induction therapy using either the DVRd regimen (Daratumumab, Bortezomib, Lenalidomide, and Dexamethasone) or the DKRd regimen (Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone).

Following induction, patients will undergo high-dose melphalan conditioning followed by autologous hematopoietic stem cell transplantation. On Day 5 after stem cell reinfusion, patients will receive anti-BCMA CAR-T cell infusion.

After CAR-T therapy, patients will enter the maintenance phase with lenalidomide monotherapy or lenalidomide in combination with bortezomib until disease progression or intolerable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 70 years; Estimated life expectancy > 12 weeks; Diagnosis of multiple myeloma confirmed by physical examination, histopathology, laboratory tests, and imaging; Liver function: ALT and AST < 3 times the upper limit of normal; Karnofsky Performance Status (KPS) score > 50%; No severe dysfunction of major organs such as the liver or heart; Willingness to undergo ASCT and CAR-T cell therapy for multiple myeloma; Ability to provide peripheral venous blood and no contraindications to leukapheresis; Ability to understand the study and sign a written informed consent voluntarily.

Exclusion Criteria:

Pregnant or lactating women, or those planning pregnancy within six months; Patients with infectious diseases, including HIV infection or active tuberculosis; Patients with active hepatitis B or C virus infection; Pre-screening indicates peripheral blood T cell transduction efficiency <10% or expansion fold <5× under CD3/CD28 co-stimulation; Patients with abnormal vital signs or unable to cooperate with the procedures; Patients with psychiatric or psychological disorders that impair compliance or assessment; Patients with a history of severe allergies or hypersensitivity, particularly to interleukin-2 (IL-2); Patients with systemic or severe local infections requiring anti-infective therapy; Patients with significant dysfunction of vital organs such as the heart, lungs, or brain; Any other condition deemed unsuitable for participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Month 6, 12, 18 and 24
  The proportion of patients achieving partial response (PR) or better according to the IMWG criteria.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Month 6, 12, 18 and 24
  Time from CAR-T infusion to disease progression or death from any cause.
Overall Survival (OS) | Month 6, 12, 18 and 24
  Time from CAR-T infusion to death from any cause.

IPD SHARING:
Plan to Share IPD: No